CLINICAL TRIAL: NCT06310499
Title: Primary or Secondary Fatal Drowning? A Registry-based Study Analysing Autopsy Reports From Patients Registered in the Danish Prehospital Drowning Data
Brief Title: Primary or Secondary Drowning
Acronym: DROWN_COD
Status: Active, not recruiting | Type: Observational
Sponsor: Prehospital Center, Region Zealand (Other)
Responsible Party: Principal Investigator, Niklas Breindahl, Principal Investigator, Prehospital Center, Region Zealand
Other Study IDs: DROWN_COD
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Drowning; Drowning; Anoxia; Drowning, Near; Drowning in Swimming Pool; Drowning; Asphyxia; Drowning/Diving/SCUBA Accident; Drowning or Immersion of Unknown Intent; Drowning and Submersion, Undetermined Intent; Drowning and Submersion While in Bath-Tub; Drowning and Submersion While in Natural Water; Drowning and Submersion Due to Sailboat Sinking; Drowning and Submersion Due to Fall Off Ship; Drowning and Submersion While in Swimming-Pool
Keywords: Drowning; Epidemiology; Danish Prehospital Drowning Data; Danish Drowning Formula; Registry; Cohort; Autopsy; Cause of death; Death certificate; Database; Denmark; Utstein
MeSH Terms: conditions — Drowning; Hypoxia; Near Drowning; Asphyxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Primary fatal drowning: These patients are registered in the Danish Register of Causes of Death, with drowning as an underlying cause of death in the death certificate.
  Interventions: Other: Drowning
- Secondary fatal drowning: These patients are registered in the Danish Register of Causes of Death, with drowning as a contributory cause of death or drowning not registered in the death certificate.
  Interventions: Other: Drowning

INTERVENTIONS:
Other: Drowning — Drowning is defined as the process of experiencing respiratory impairment from submersion or immersion in liquid.

SUMMARY:
According to WHO's rules, any death certificate must state the underlying cause of death and contributory causes of death may also be stated.

Differentiating between primary and secondary drowning is difficult, as information preceding the drowning incident is rarely available. Yet, knowing the most frequent causes of secondary drowning may provide useful information to healthcare professionals working in prehospital Emergency Medical Services, as this may affect prehospital treatment.

DETAILED DESCRIPTION:
The annual death statistics are based solely on the underlying cause of death, that is the disease or condition which started the process that led to death. The conditions that directly caused the death are also to be stated by the physician on the death certificate and may be included in the statistics. In research projects, data on those contributory causes of death may be drawn from the register. It is now the medical doctor who has verified the death and issued the death certificate indicating the underlying and contributory causes of death, who also classifies these causes in accordance with ICD-10 and fills in the coded data on the electronic death certificate. The Danish Register of Causes of Death is, thus, updated without central validation of the classification and relies entirely on the coding done by individual physicians.

This study aims to characterise fatal drowning incidents as primary or secondary drownings and report the frequencies of secondary drowning causes.

ELIGIBILITY:
Inclusion Criteria:

* All drowning patients registered in the Danish Prehospital Drowning Data AND
* Having a fatal outcome within 30 days after the drowning incident AND
* Having a valid civil registration number in the Danish Prehospital Drowning Data
* Being able to link data from the Danish Register of Causes of Death

Exclusion Criteria:

* Patients alive 30 days after the drowning incident
* Patients with an invalid civil registration number in the Danish Prehospital Drowning Data
* Patients where data cannot be retrieved from the Danish Register of Causes of Death

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Danish Prehospital Drowning Data reports prehospital data on patients with fatal and non-fatal drowning treated by the Emergency Medical Services in Denmark since 2016. Drowning incidents are identified from the Danish Prehospital Electronic Medical Record using the Danish Drowning Formula and extensive manual validation. Data is extracted following the revised USFD. The patients' unique civil registration number enable linkage with the Civil Personal Register to obtain data on 30-day survival and differentiate between fatal and non-fatal drowning incidents
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Autopsy rate | Data is extracted on patients registered in the Danish Prehospital Drowning Data from 2016-2023.
  Calculated as the number of autopsy reports divided by the number of fatal drowning incidents registered in the Danish Prehospital Drowning Data.
Primary fatal drowning rate | Data is extracted on patients registered in the Danish Prehospital Drowning Data from 2016-2023.
  Calculated as the number of autopsy reports stating drowning as the underlying cause of death divided by the number of fatal drowning incidents registered in the Danish Prehospital Drowning Data.
Secondary fatal drowning rate | Data is extracted on patients registered in the Danish Prehospital Drowning Data from 2016-2023.
  Calculated as the number of autopsy reports stating drowning as the contributory cause of death OR not stating drowning as a contributory cause of death divided by the number of fatal drowning incidents registered in the Danish Prehospital Drowning Data.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Collatz Christensen, Ass. Prof., Study Director — Prehospital Center, Region Zealand
Locations (1):
- Prehospital Center, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No
The data are available upon reasonable request from researchers after application to the corresponding author, provided the necessary approvals are obtained from the relevant authorities.

REFERENCES:
- [Background] Breindahl N, Wolthers SA, Jensen TW, Holgersen MG, Blomberg SNF, Steinmetz J, Christensen HC; Danish Cardiac Arrest Group. Danish Drowning Formula for identification of out-of-hospital cardiac arrest from drowning. Am J Emerg Med. 2023 Nov;73:55-62. doi: 10.1016/j.ajem.2023.08.024. Epub 2023 Aug 15. PMID 37619443
- [Background] Helweg-Larsen K. The Danish Register of Causes of Death. Scand J Public Health. 2011 Jul;39(7 Suppl):26-9. doi: 10.1177/1403494811399958. PMID 21775346